CLINICAL TRIAL: NCT07225686
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Maridebart Cafraglutide in Adult Participants With Obstructive Sleep Apnea on Positive Airway Pressure Therapy and Living With Overweight or Obesity
Brief Title: Maridebart Cafraglutide Versus Placebo in Adult Participants With Obstructive Sleep Apnea on Positive Airway Pressure Therapy
Acronym: MARITIME-OSA-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230225
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Obstructive Sleep Apnea
Keywords: MariTide; Maridebart Cafraglutide; AMG 133; Obesity
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maridebart Cafraglutide (Experimental): Participants will receive maridebart cafraglutide subcutaneously (SC).
  Interventions: Drug: Maridebart cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart cafraglutide — Participants will receive maridebart cafraglutide as SC injections.
  Other Names: AMG 133
  Arms: Maridebart Cafraglutide
Drug: Placebo — Participants will receive placebo SC.
  Arms: Placebo

SUMMARY:
This Phase 3 clinical trial is designed to evaluate the efficacy and safety of maridebart cafraglutide compared to placebo over a 52-week period in adults with obstructive sleep apnea (OSA) who are receiving positive airway pressure (PAP) therapy and are living with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* AHI ≥ 15 on polysomnography at day 1 before randomization.
* BMI ≥ 27 kg/m^2 at screening.
* History of at least 1 unsuccessful attempt at weight loss by diet and exercise.
* On positive airway pressure (PAP) therapy for at least 3 consecutive months before screening and plan to continue PAP therapy during the trial.

Exclusion Criteria:

* Had any previous or planned upper airway surgery for sleep apnea or major ear, nose, or throat surgery.
* Significant craniofacial abnormalities that may affect breathing at screening.
* Diagnosis of Central Apnea with % of central apneas/hypopneas ≥ 50%, and/or diagnosis of Cheyne Stokes Respiration.
* Active device treatment of obstructive sleep apnea other than PAP therapy (eg, oral appliances), or other treatments, that in the opinion of the investigator, may interfere with trial outcomes, unless willing to stop treatment at screening and throughout the trial.
* Respiratory diseases such as obesity hypoventilation syndrome or daytime hypercapnia, or neuromuscular diseases such as myasthenia gravis or other conditions that could interfere with the results of the trial in the opinion of the investigator.
* Have personal circumstances or job-related responsibilities that prevent a 7-day PAP withdrawal before polysomnography testing during the course of the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2028-09-13 (Estimated)

PRIMARY OUTCOMES:
Change in AHI from baseline at week 52 | At Week 52

SECONDARY OUTCOMES:
Percentage Change in AHI from baseline at week 52 | At Week 52
Participants Achieving ≥ 50% AHI Reduction from baseline at week 52 | At Week 52
Participants Achieving AHI < 5 or AHI 5 to 14 with Epworth Sleepiness Scale (ESS) ≤ 10 from baseline at week 52 | At Week 52
Percentage Change in Body Weight from baseline at Week 52 | At Week 52
Change in Sleep Apnea-specific Hypoxic Burden (SASHB) from baseline at Week 52 | At Week 52
Change in High Sensitivity C-reactive Protein (hs-CRP) from baseline at Week 52 | At Week 52
Change in Systolic Blood Pressure from baseline at Week 48 | At Week 48
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Sleep-related Impairment 8a Score from baseline at Week 52 | At Week 52

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (11):
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Teradan Clinical Trials, Brandon, Florida
  - Destiny Research Center, Palmetto Bay, Florida
  - Clinical Research Center Of Florida, Pompano Beach, Florida
  - Basil Clinical, Laurelton, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - FutureSearch Trials of Neurology, Austin, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Australia (2):
  - Woolcock Institute of Medical Research, Macquarie Park, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
- Canada (2):
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Wharton Medical Clinic, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com